CLINICAL TRIAL: NCT03367091
Title: Energy Consumption and Cardiorespiratory Load During Overground Gait Training With a Wearable Exoskeleton After Stroke: the Effect of the Level of Swing Assistance
Brief Title: Energy Consumption and Cardiorespiratory Load During Overground Gait Training With a Wearable Exoskeleton After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisational/Recruitment Issues
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Nina Lefeber, Doctoral Researcher, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EKSO STUDY I
Record Dates: First submitted 2017-11-30; First posted 2017-12-08 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Stroke
Keywords: Wearable Exoskeleton; Stroke; Energy Consumption; Cardiorespiratory Load
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ekso GT gait training (Experimental): Participants will be measured during three Ekso GT gait trainings:
  * 20-minute Ekso GT gait training with high swing assistance
  * 20-minute Ekso GT gait training with neutral swing assistance
  * 20-minute Ekso GT gait training with high swing resistance.
  Each training will be performed on a separate day in a randomized order (within one week and controlled for time of day).
  Interventions: Other: Ekso GT gait training with high swing assistance; Other: Ekso GT gait training with neutral swing assistance; Other: Ekso GT gait training with high swing resistance

INTERVENTIONS:
Other: Ekso GT gait training with high swing assistance — Participant will walk for 20-minutes in the Ekso GT SmartAssist with the swing assistance set at "high assistance"
Other: Ekso GT gait training with neutral swing assistance — Participant will walk for 20-minutes in the Ekso GT SmartAssist with the swing assistance set at "neutral"
Other: Ekso GT gait training with high swing resistance — Participant will walk for 20-minutes in the Ekso GT SmartAssist with the swing assistance set at "high resistance"

SUMMARY:
To investigate acute metabolic and cardiorespiratory responses during overground gait training with a wearable exoskeleton in persons after stroke

DETAILED DESCRIPTION:
RESEARCH AIMS:

* To investigate the effect of the level of swing assistance on the acute metabolic and cardiorespiratory responses during overground gait training with a wearable exoskeleton in persons after stroke
* To investigate if there is an interaction-effect between the level of swing assistance and the duration of walking
* To compare the exercise intensity to aerobic training recommendations

STUDY DESIGN: An experimental, 1-group trial with randomized crossover design.

PATIENT RECRUITMENT: Participants will be recruited at the AZ Herentals (Herentals, Belgium).

LOCATION: The trial will be conducted at the REVAlution Center (Herentals, Belgium).

ELIGIBILITY CRITERIA: See section "Eligibility"

PROCEDURES: Before the start of the study, informed consent and baseline patient characteristics will be collected. Next, participants will be measured during three training sessions with the Ekso GT SmartAssist:

* 20-minute training with high swing assistance
* 20-minute training with neutral swing assistance
* 20-minute training with high swing resistance

Trainings will be performed on a separate day in a randomized order (within one week and controlled for time of day).

Following settings will be used in all three conditions: sitting program ("Min lean"); standing program ("Auto lean"); step initiation program ("ProStep+"), training mode ("Off"), SmartAssist option ("2Free"); and stance support ("Low"). The level of stance support and swing assistance will be set symmetrically for the affected and non-affected side.

During training, participants will walk back and forth at a self-selected walking speed in a 30m hall way using a cane at the non-affected side.

Prior to the experimental conditions, participants will have had three training sessions in the Ekso GT.

RESTRICTIONS & PROHIBITIONS: Participants will be instructed to not consume food, alcohol, caffeine or nicotine at least 3h prior to the intervention. Usual medication intake will be allowed with small amounts of water.

MATERIALS: The Ekso GT robotic exoskeleton with SmartAssist (Ekso Bionics Inc., USA) will be used during the overground training sessions.

A flexible facemask (adult facemask, small/medium, Cortex, Germany), lightweight chest carrying gas analysis system (Metamax 3B, Cortex, Germany) and Bluetooth heart rate belt (Polar H7, Polar Electro, Finland) will be used to measure metabolic and cardiorespiratory parameters. At the start of each measurement, gas (room air and reference gas (17.4% O2 and 5.1% CO2)) and volume (3L syringe) calibrations of the breath-by-breath gas analysis system will be performed in accordance with the manufacturer's instructions.

OUTCOMES: See section "Outcome Measures"

DATA-ANALYSES: Descriptive statistics will be calculated for baseline patient characteristics. To investigate the effect of level of swing assistance and duration, a repeated measures ANOVA (within factor duration and within factor assistance level) will be conducted (interaction-effect time x duration, main effect assistance level and main effect duration). In case of significant differences, posthoc analyses will be interpreted. The walking speed will be considered as a covariate in the ANOVA analysis (in case significant different between conditions). Significance level will be set at 5%.

ELIGIBILITY:
Included will be persons who

* Had a stroke
* Cannot walk independently or can walk independently on level ground, but still require help on stairs, slopes or uneven surfaces (FAC 0 - 4)

Excluded will be persons who

* Can walk independently on level ground, stairs, slopes and uneven surfaces (FAC 5)
* Have musculoskeletal problems (other than stroke) affecting the ability to walk
* Have concurrent pulmonary diseases (e.g. asthma)
* Have unstable cardiovascular conditions
* Have concurrent neurological diseases (e.g. Parkinson's Disease)
* Have communicative and/or cognitive problems affecting the ability to understand or follow instructions
* Present contra-indications for using the Ekso GT (according to manufacturer's instructions)

  * Severe concurrent medical diseases (infections, circulatory, heart or lung, pressure sores)
  * Severe spasticity (Ashworth 4)
  * Range of motion restrictions that would prevent a patient from achieving normal, reciprocal gait pattern, or would restrict a patient from completing normal sit-to-stand or stand-to-sit transitions

    * Bilateral hip flexion < 110°
    * Knee flexion contracture > 12°
    * Inability to achieve 0° neutral angle dorsiflexion with knee flexion ≤ 12°
  * Weight ≥ 100 kg
  * Hip width < 35.8 cm or > 45.6 cm
  * Upper leg length < 51 cm or > 61.4 cm
  * Lower leg length < 48 cm or > 63.4 cm
  * Upper leg length discrepancy > 0.5 inch (1.3 cm)
  * Lower leg length discrepancy > 0.75 inch (1.9 cm)
  * Unstable spine, unhealed limbs or pelvic fractures
  * Unhealthy bone density
  * Heterotopic ossification
  * Significant contractures
  * Elbows and shoulders are unable to support crutches, walker or cane
  * Psychiatric or cognitive situations that may interfere with proper operation of the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Net oxygen cost (OC, ml/kg/m) at minute 5 of walking | Minute 5 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net oxygen cost (OC, ml/kg/m) at minute 10 of walking | Minute 10 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net oxygen cost (OC, ml/kg/m) at minute 15 of walking | Minute 15 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net oxygen cost (OC, ml/kg/m) at minute 20 of walking | Minute 20 of 20-minute walking period
  Net oxygen consumption (oxygen consumption (ml/kg/min) during walking minus during rest) divided by the walking speed (m/min)
Net heart rate (HR, beats/min) at minute 5 of walking | Minute 5 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net heart rate (HR, beats/min) at minute 10 of walking | Minute 10 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net heart rate (HR, beats/min) at minute 15 of walking | Minute 15 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net heart rate (HR, beats/min) at minute 20 of walking | Minute 20 of 20-minute walking period
  Heart rate during walking (beats/min) minus resting heart rate
Net minute ventilation (VE, L/min) at minute 5 of walking | Minute 5 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest
Net minute ventilation (VE, L/min) at minute 10 of walking | Minute 10 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest
Net minute ventilation (VE, L/min) at minute 15 of walking | Minute 15 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest
Net minute ventilation (VE, L/min) at minute 20 of walking | Minute 20 of 20-minute walking period
  The amount of air in- or exhaled per minute (L/min) during walking minus during rest

SECONDARY OUTCOMES:
Net Rating of Perceived Exertion (RPE, 6-20) at minute 5 of walking | Minute 5 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest
Net Rating of Perceived Exertion (RPE, 6-20) at minute 10 of walking | Minute 10 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest
Net Rating of Perceived Exertion (RPE, 6-20) at minute 15 of walking | Minute 15 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest
Net Rating of Perceived Exertion (RPE, 6-20) at minute 20 of walking | Minute 20 of 20-minute walking period
  Rating of perceived effort, strain and/or fatigue during walking, pointed on a 15-point Borg scale (6-20) during walking minus during rest
Percentage maximal heart rate (%HRmax) at minute 5 of walking | Minute 5 of 20-minute walking period
  Heart rate divided by predicted maximum heart rate.
Percentage maximal heart rate (%HRmax) at minute 10 of walking | Minute 10 of 20-minute walking period
  Heart rate divided by predicted maximum heart rate.
Percentage maximal heart rate (%HRmax) at minute 15 of walking | Minute 15 of 20-minute walking period
  Heart rate divided by predicted maximum heart rate.
Percentage maximal heart rate (%HRmax) at minute 20 of walking | Minute 20 of 20-minute walking period
  Heart rate divided by predicted maximum heart rate.
Percentage heart rate reserve (%HRR) at minute 5 of walking | Minute 5 of 20-minute walking period
  Heart rate during walking minus during rest divided by predicted heart rate reserve (i.e. predicted maximum heart rate minus resting heart rate)
Percentage heart rate reserve (%HRR) at minute 10 of walking | Minute 10 of 20-minute walking period
  Heart rate during walking minus during rest divided by predicted heart rate reserve (i.e. predicted maximum heart rate minus resting heart rate)
Percentage heart rate reserve (%HRR) at minute 15 of walking | Minute 15 of 20-minute walking period
  Heart rate during walking minus during rest divided by predicted heart rate reserve (i.e. predicted maximum heart rate minus resting heart rate)
Percentage heart rate reserve (%HRR) at minute 20 of walking | Minute 20 of 20-minute walking period
  Heart rate during walking minus during rest divided by predicted heart rate reserve (i.e. predicted maximum heart rate minus resting heart rate)
Metabolic Equivalent of Task (MET) at minute 5 of walking | Minute 5 of 20-minute walking period
  Expression of the intensity of walking defined as the oxygen consumption (ml/kg/min) during walking divided by the oxygen consumption (ml/kg/min) in rest
Metabolic Equivalent of Task (MET) at minute 10 of walking | Minute 10 of 20-minute walking period
  Expression of the intensity of walking defined as the oxygen consumption (ml/kg/min) during walking divided by the oxygen consumption (ml/kg/min) in rest
Metabolic Equivalent of Task (MET) at minute 15 of walking | Minute 15 of 20-minute walking period
  Expression of the intensity of walking defined as the oxygen consumption (ml/kg/min) during walking divided by the oxygen consumption (ml/kg/min) in rest
Metabolic Equivalent of Task (MET) at minute 20 of walking | Minute 20 of 20-minute walking period
  Expression of the intensity of walking defined as the oxygen consumption (ml/kg/min) during walking divided by the oxygen consumption (ml/kg/min) in rest

OTHER OUTCOMES:
Walking speed (m/min) at minute 5 of walking | Minute 5 of 20-minute walking period
  The distance (meters) walked per minute
Walking speed (m/min) at minute 10 of walking | Minute 10 of 20-minute walking period
  The distance (meters) walked per minute
Walking speed (m/min) at minute 15 of walking | Minute 15 of 20-minute walking period
  The distance (meters) walked per minute
Walking speed (m/min) at minute 20 of walking | Minute 20 of 20-minute walking period
  The distance (meters) walked per minute

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kerckhofs, Prof, PhD, Study Chair — Vrije Universiteit Brussel; Eva Swinnen, Prof, PhD, Study Director — Vrije Universiteit Brussel; Nina Lefeber, PhD student, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- REVAlution center, Herentals, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided